CLINICAL TRIAL: NCT04963842
Title: Combining the Effects of Avoiding the Consumption of Packaged Food and Promoting the Use of Bioplastic Food Packaging on the Body Burden of Plasticizers in Young Women: A Pilot Cross-over Study
Brief Title: Investigation on the Benefits of Avoiding Conventional Food Packaging and Promoting Bioplastic Food Packaging
Acronym: BIOFOODPACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Konstantinos Makris, Associate Professor of Environmental Health, Cyprus University of Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BIOFOODPACK
Record Dates: First submitted 2021-06-18; First posted 2021-07-15 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional phase (use of conventional food packaging material) (No Intervention): During the conventional phase, participants are asked to maintain their usual habits for 5 days.
- Intervention phase (use of bio-plastic and no plastic food packaging material) (Experimental): During the 5-day long intervention period, all participants will be asked to: i) refrain from packaged (cans, plastic, paper) ready to consume foods, and foods from take away/delivery/fast food and ii) use the bio-based food packaging material to package their food.
  Interventions: Behavioral: Use of bio-plastic food packaging material and avoidance of plastic food packaging material

INTERVENTIONS:
Behavioral: Use of bio-plastic food packaging material and avoidance of plastic food packaging material — The bio-plastic food packaging material will be used by the study participants for 5 days and no plastic packaged food will be consumed.
  Arms: Intervention phase (use of bio-plastic and no plastic food packaging material)

SUMMARY:
A trial study was proposed as part of the project "Biocomposite Packaging for Active Preservation of Food" (acronym BIOFOODPACK) that has been funded by the M-ERA.Net Call 2016. A crossover trial with a behavioral intervention study will be conducted. The behavioural intervention treatment consists of: i) avoiding the consumption of packaged (cans, plastic, paper) ready to consume foods, and foods from take away/delivery/fast food, and ii) using the proposed bio-based packaging material to package foods ready for consumption; this bio-based packaging material (Silvex Ltd, Portugal) does not contain plasticizers, it is biodegradable and made out of plant-based materials (corn, starch, etc.). The objectives of this study are:

1. To describe the body burden of plasticizers for women aged 18-40 years systematically adopting the intervention treatment package during the 5-day period.
2. To assess the diurnal variability of the plasticizers, based on regular daily activities of the young adult women.

DETAILED DESCRIPTION:
The duration of this study will be 12 days; the intervention period will last for 5-days, followed by the 2-day wash out and then another 5-day period for the conventional period (as usual) (Figure 1). During the 5-day long intervention period, all participants will be asked to: i) refrain from packaged (cans, plastic, paper) ready to consume foods, and foods from take away/delivery/fast food and ii) use the bio-based food packaging material to package their food.

The participants will be randomly allocated to the treatment period or the conventional period (as usual scenario) for 5 days, each and following a washout period of 2 days, they will use the biodegradable food packaging material and no plastic packaging for their ready to eat foods for the next 5 days.

A baseline questionnaire will be used to collect information on demographic characteristics, individual habits, diet and non-dietary potential endocrine-disruptive chemicals exposures, while a diary will be used daily by participants so that they report the time for consumption of packaged food/drinks, for use of personal care products and for other activities like handwashing and use of microwave. Both the baseline questionnaire and diary will be developed online using the REDCap platform. Participants will provide us with an informed consent that they will strictly follow the protocol in both phases.

Standardized methodologies to quantify endocrine-disruptive chemicals (bisphenols, free and total) in urine samples and in packaged food using standardized protocols will be used. Urine samples will be analyzed at the Water and Health laboratory for plasticizers (bisphenols both free and total forms) using established human biomonitoring methods. The methods for the plasticizer compounds will be those used by the U.S. CDC. Standardized measurements for metabolomics and cortisol will also take place.

ELIGIBILITY:
Inclusion Criteria:

* Ηealthy young women at the age of 18-40 years old, who reside in Cyprus at least the last five years. Also, subjects will be included if they routinely consume food previously packaged in plastic packaging materials/boxes

Exclusion Criteria:

* Women with medical history, such as those taking medication for any chronic disease such as asthma, type I diabetes and those who systematically don't use or buy plastic packaged food.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Urinary plasticizers levels during the study period | 10 days
  Assess if plasticizers levels such as bisphenols (free and total) differ between the intervention phase and the conventional phase. Plasticizers will be measured in spot urine samples of day 1 and 5 of each phase using GC-MS/MS methodology.
Diurnal variability of urinary plasticizers levels during the study period | 10 days
  Assess the diurnal variability of plasticizers, based on regular daily activities of the young adult women that will be recorded in the diary and the plasticizers levels in the spot urine samples taken on day 1 and day 5 of each phase. Plasticizers will be measured using GC-MS/MS methodology.

SECONDARY OUTCOMES:
Diurnal variability of urinary cortisol levels during the study period | 10 days
  Assess the diurnal variability of cortisol, based on regular daily activities of the young adult women that will be recorded in the diary and the cortisol levels in the spot urine samples taken on day 1 and day 5 of each phase. Cortisol will be measured using GC-MS/MS methodology.
Differentiated metabolite change (fold change) for metabolomics platform-based profiles in two study periods | 10 days
  Untargeted GC-MS metabolomics analysis

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Makris, PhD, Principal Investigator — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Upon publication, anonymized data will be shared
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Upon publication
Access Criteria: Open Access